CLINICAL TRIAL: NCT00668980
Title: The Constitution of Symbolic Representation in Young Children With Down Syndrome
Brief Title: Symbolic Representation in Young Children With Down Syndrome
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Suelly Cecilia Olivan Limongi, University of Sao Paulo
Other Study IDs: 06/50842-4
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Down Syndrome
Keywords: Down syndrome; symbolic representation; gestures; expressive language development
MeSH Terms: conditions — Down Syndrome; Gestures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: 20 infants with Down syndrome
- Control Group: 15 typically developing children

SUMMARY:
The aim of this study is to characterize the process of constitution of symbolic representation in infants with Down syndrome, as well as to investigate the relationship between gestures and the emergence of oral language. The investigators hypothesis is that children with Down syndrome could present difficulties during the constitution of symbolic representation that may be related to later deficits on expressive language, generally observed in these children.

DETAILED DESCRIPTION:
According to the Genetic Epistemology, language development is directly related to cognitive construction. Such relationship is clearly observed after the constitution of representation that allows one individual to express his or her thinking through language.

ELIGIBILITY:
Inclusion Criteria for Study Group:

* genetic diagnosis of Down Syndrome
* be at the 4th stage of sensorimotor period at the initial assessment
* good health conditions
* good results on audiologic evaluation
* pediatric and ear, nose and throat periodic check ups.

Inclusion Criteria for Control Group:

* good health conditions
* be at the 4th stage of sensorimotor period at the initial assessment
* pediatric and ear, nose and throat periodic check ups.

Exclusion Criteria for all groups:

* submission to long term hospitalizations due to heart diseases and major respiratory airway infections, that may interfere in the child's global development
* presence of visual or auditory important deficits
* historic of prematurely and/or low birth weight

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Group - children with Down syndrome that attend speech-language therapy at the Speech Language Pathology Laboratory in Syndromes and Sensorimotor Deficits of the School of Medicine of the University of São Paulo or from the Association of Parents and Friends of Exceptional children of São José dos Campos.
  Control Group
  - typically developing children followed up in the Pediatrics Ambulatory of the University's Hospital and/or being assisted in the University' Hospital Nursery School.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Performance on monthly assessments administered after the initial evaluation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Suelly CO Limongi, PhD., Study Chair — University of Sao Paulo; Fabiola C Flabiano, PhD. student, Principal Investigator — University of Sao Paulo
Locations (3):
- Brazil (3):
  - APAE Sao José dos Campos, São José dos Campos, São Paulo
  - University Hospital, São Paulo, São Paulo
  - University of Sao Paulo - School of Medicine - Department of Physiotherapy, Communication Sciences and Disorders, Occupational Therapy, São Paulo, São Paulo